CLINICAL TRIAL: NCT04767607
Title: International Peace Maternity and Child Health Hospital (IPMCH) Affiliated to School of Medicine, Shanghai Jiaotong University, Shanghai, China
Brief Title: Study of Prediction of Ovarian Reserve in Yong Breast Cancer Patients Treated With Chemotherapy
Status: Completed | Type: Observational
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Collaborators: School of Biomedical Engineering, Shanghai Jiao Tong University (Unknown)
Responsible Party: Principal Investigator, Dongmei Lai, Principal Investigator, International Peace Maternity and Child Health Hospital
Other Study IDs: GFY202001
Record Dates: First submitted 2021-01-26; First posted 2021-02-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Chemotherapy; ovarian reserve
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer plus chemotherapy: Patients of the group will receive chemotherapy treatment.
- Breast cancer without chemotherapy: Patients of the group will not receive chemotherapy treatment.

SUMMARY:
The purpose of this study is to predict the ovarian reserve, especially premature ovarian insufficient (POI), in young breast cancer patients during chemotherapy treatment using ultrasensitive anti-Müllerian hormone (AMH) detection method.

DETAILED DESCRIPTION:
Young breast cancer women are often treated with adjuvant chemotherapy and neoadjuvant chemotherapy regiments include cyclophosphamide, anthracyclines and a taxane. These treatments can adversely affect ovarian function across the lifespan, causing premature menopause, infertility, and POI. AMH is currently the most robust marker of prediction of ovarian injury in cancer patients during chemotherapy in compare with other sexual hormone marker (such as follicle stimulating hormone (FSH), inhibin B) and ovarian volume, and is a more convenient way of prediction of ovarian reserve compare antral follicle count (AFC). But most of the patients' AMH levels become undetectable (using common AMH kits) after several cycle of chemotherapy, and some of these patients' AMH levels will maintained at a low level after chemotherapy, while others will recover. Using the ultrasensitive AMH detection method is expected to accurately assess the ovarian reserve during the chemotherapy treatment, predicting the risk of ovarian failure, and providing patients with ovarian and fertility function protection recommendations, such as using GnRHa regents during treatment and providing assisted reproductive technology consultants.

ELIGIBILITY:
Inclusion Criteria:

1. Female 18-50 years.
2. Suffering from breast cancer.
3. Treated with adjuvant or neoadjuvant chemotherapy.
4. Having regular menstrual cycle before chemotherapy.

Exclusion Criteria:

1. Bilateral oophorectomy or ovarian irradiation before enrollment.
2. Prior chemotherapy.
3. Oral contraceptives before enrollment.
4. Pregnancy or lactation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 premenopausal breast cancer female patients of age 18-50 treated in the International Peace Maternity and Child Health Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the trend of anti-Müllerian hormone (AMH) level at chemotherapy process and post-chemotherapy in breast cancer patients. | 1 year.
  Serum anti-Müllerian hormone (AMH) concentration can be measured on any day during the menstrual cycle. Serum AMH will be measured at each chemotherapy administration and 1 year post-chemotherapy.

SECONDARY OUTCOMES:
To evaluate the trend of Follicle-Stimulating Hormone (FSH) level at chemotherapy process and post-chemotherapy in breast cancer patients. | 1 year.
  Serm FSH concentration will be measured at each chemotherapy process and 1 year post-chemotherapy.

OTHER OUTCOMES:
Number of participants with chemotherapy-induced amenorrhoea/oligomenorrhea and recovery rate of menses during chemotherapy process and 1 year post-chemotherapy treatment. | 1 year.
  Disappearance and reappearance of two consecutive menstrual periods within 21 to 35 days during chemotherapy treatment and 1 year post-chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Lai, M.D., Principal Investigator — The International Peace Maternity and Child Health Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- The International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The public can require the data and protocol from clinicaltrials.gov posted by investigator.
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: Public
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Dezellus A, Barriere P, Campone M, Lemanski C, Vanlemmens L, Mignot L, Delozier T, Levy C, Bendavid C, Debled M, Bachelot T, Jouannaud C, Loustalot C, Mouret-Reynier MA, Gallais-Umbert A, Masson D, Freour T. Prospective evaluation of serum anti-Mullerian hormone dynamics in 250 women of reproductive age treated with chemotherapy for breast cancer. Eur J Cancer. 2017 Jul;79:72-80. doi: 10.1016/j.ejca.2017.03.035. Epub 2017 Apr 29. PMID 28463758
- [Background] Freour T, Barriere P, Masson D. Anti-mullerian hormone levels and evolution in women of reproductive age with breast cancer treated with chemotherapy. Eur J Cancer. 2017 Mar;74:1-8. doi: 10.1016/j.ejca.2016.12.008. Epub 2017 Jan 28. PMID 28135602
- [Background] Lie Fong S, Lugtenburg PJ, Schipper I, Themmen AP, de Jong FH, Sonneveld P, Laven JS. Anti-mullerian hormone as a marker of ovarian function in women after chemotherapy and radiotherapy for haematological malignancies. Hum Reprod. 2008 Mar;23(3):674-8. doi: 10.1093/humrep/dem392. Epub 2008 Jan 23. PMID 18216040